CLINICAL TRIAL: NCT06641518
Title: Effectiveness of Transcutaneous Electrical Nerve Stimulation Combined With Task-Related Training on Upper Limb Function in Subacute Hemiparetic Stroke Patients
Brief Title: Effectiveness of TENs Combined With Task-Related Training on Upper Limb Function in Subacute Hemiparetic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Songsuda Roongsaiwatana, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COA.MURA2021/831
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Upper Limb Function in Subacute Hemiparetic Stroke Patients
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): Transcutaneous Electrical Nerve Stimulation (TENS) was applied to the brachial plexus at the supraclavicular fossa (Erb's point) and to the radial nerve between the biceps and triceps in the spiral groove. The frequency was set at 10 Hz, and the intensity was adjusted to a level that elicited sensation without causing pain or muscle twitching, for a duration of 45 minutes, five days a week, totaling 20 sessions over four weeks, combined with standard upper extremity conservative occupational therapy training.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Sham TENS (Sham Comparator): Transcutaneous Electrical Nerve Stimulation (TENS) on the affected arm according to the same treatment protocol as above; however, the device was not turned on, and no electrical current was delivered (Placebo).
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — a therapeutic modality employing electric current to relieve pain by activating peripheral nerves. The evolution of TENS units alongside technological advancements has led to user-friendly interfaces and enhanced portability, with units now small enough to be carried in a pocket.

SUMMARY:
To study the effectiveness of transcutaneous electrical nerve stimulation (TENS) combined with occupational therapy on restoring the function of the weakened limb in subacute stroke patients.

DETAILED DESCRIPTION:
To study the effectiveness of transcutaneous electrical nerve stimulation (TENS) combined with occupational therapy on restoring the function of the weakened limb in subacute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a first-ever stroke, presenting with unilateral weakness and accompanying arm weakness, in the subacute phase (2 weeks - 6 months).
* Able to follow commands and cooperate in an active training program.
* Patients must consent to participate in the research project by signing a consent form.
* Aged between 18 and 80 years.
* Exhibiting mild to moderate muscle spasticity (Modified Ashworth Scale < 3).

Exclusion Criteria:

* Patients with other neurological disorders, such as traumatic brain injury or spinal cord injury, or those experiencing severe complications from treatment.
* Unable to tolerate the use of TENS.
* Contraindications for using TENS, such as having a pacemaker or infected skin lesions.
* Unstable or uncontrolled vital signs or other comorbidities.
* Communication difficulties that prevent following commands or cooperating in training.
* Participants who refuse or withdraw from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of upper extremity scores (FMA-UE) | baseline, 2 weeks, 4 weeks, and 8 weeks post-intervention.
  a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia

SECONDARY OUTCOMES:
Wolf motor function test (WMFT) | baseline, 2 weeks, 4 weeks, and 8 weeks post-intervention.
  measures upper extremity (UE) motor abilities
Box and block test (BBT) | baseline, 2 weeks, 4 weeks, and 8 weeks post-intervention.
  measures unilateral gross manual dexterity
Modified functional reach test (FRT) | baseline, 2 weeks, 4 weeks, and 8 weeks post-intervention.
  a patient's stability by measuring the maximum distance an individual can reach forward while standing in a fixed position.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical medicine and rehabilitation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrico C, Westgate PM, Salmon Powell E, Chelette KC, Nichols L, Pettigrew LC, Sawaki L. Nerve Stimulation Enhances Task-Oriented Training for Moderate-to-Severe Hemiparesis 3-12 Months After Stroke: A Randomized Trial. Am J Phys Med Rehabil. 2018 Nov;97(11):808-815. doi: 10.1097/PHM.0000000000000971. PMID 29794530